CLINICAL TRIAL: NCT01859871
Title: Evaluation of a Culturally Competent Website on Living Kidney Donation for Hispanics
Brief Title: Evaluation of a Website on Living Kidney Donation for Hispanics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Elisa Gordon, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R39OT22059
Record Dates: First submitted 2013-05-20; First posted 2013-05-22 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: End Stage Kidney Disease
Keywords: Living kidney donation; End-stage renal disease; Latinos; Undocumented Immigrants; Bilingual; Spanish; Website; Dialysis; Hispanics; Transplantation
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Arm (No Intervention): Study participants will take the self-administered pre-test and receive the standard of care. After taking the pre-test, control arm participants will be done with study participation for that day and will attend the transplant center's education sessions. All participants will receive a letter and follow-up call at about two weeks later to schedule the final survey. They will take a final survey via telephone about 3 weeks later. The final survey includes the same topics as the pre-test. They will receive a thank you letter and gift card by mail after completing the final survey.
- Website Intervention (Experimental): Navigate website plus standard of care
  Interventions: Behavioral: Website Intervention

INTERVENTIONS:
Behavioral: Website Intervention — Study participants will take the self-administered pre-test in the intervention arm and will be introduced to the website to inform the public of various topics concerning end-stage kidney disease and kidney transplantation. Few websites about transplantation are tailored to potential Hispanic kidney transplant candidates or the Hispanic community. This website is designed to fill the void and be an effective bilingual web-based educational resource targeted to Hispanic patients and public which can serve as a culturally competent tool to enhance knowledge and attitudes about living kidney donation.
  Arms: Website Intervention

SUMMARY:
The purpose of this study is to increase understanding about living kidney donation (LKD) among Hispanic/Latino patients and public by increasing knowledge and positive attitudes about LKD. Improving Hispanics' understanding about LKD will ensure that Hispanic patients and public are fully informed of the treatment options for End Stage Kidney Disease.

DETAILED DESCRIPTION:
The shortage of kidneys for transplantation, and ethnic disparities in living kidney donation rates are major public health problems. Hispanics need more kidney transplants, yet receive fewer living donor kidney transplants than they need. Factors known to contribute to Hispanics' low rates of living donation kidney transplantation include cultural beliefs, lack of knowledge, and negative attitudes about living kidney donation. Web-based interventions are promising as Hispanics are using the Internet at increasingly greater rates. However, few websites about transplantation are tailored to potential Hispanic kidney transplant candidates or the Hispanic community. This study aims to develop, test, and evaluate the effectiveness of a bilingual web-based educational resource targeted to Hispanic patients and the public, which can serve as a low-cost, convenient, and culturally competent tool to enhance knowledge about living kidney donation. Improving Hispanics' understanding about living kidney donation will promote their autonomy and self-determination by helping to ensure that Hispanic patients and public are fully informed of the treatment options for end-stage kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥ 18 years)
* Hispanics/Latinos
* ESRD patients who are scheduled to attend each participating transplant center's education sessions. Sessions mark the first phase of evaluation in order for patients to get wait listed for a transplant or for others to become a living kidney donor.
* Family and friends who accompany patients to the transplant center.
* Identification as Hispanic/Latino.
* Ability to come to Northwestern 3 hours prior to the scheduled education session.
* Ability to read. Reading ability will be assessed using the 5-point Likert scale question validated in English and Spanish:13 "How often do you need to have someone help you when you read instructions, pamphlets, or other written material from your doctor or pharmacy?" People will be included if they reply 1-Never or 2-Rarely.

Exclusion Criteria:

* Non-identification as Hispanic/Latino.
* Inability to come to Northwestern 3 hours prior to the scheduled education session.
* Individuals who are not able to read Spanish or English. People will be excluded if they reply 3-Sometimes, 4-Often, and 5-Always to the question, "How often do you need to have someone help you when you read instructions, pamphlets, or other written material from your doctor or pharmacy?" .

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2013-05; Primary Completion 2015-02 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Knowledge about Living Kidney Donation | 3 weeks
  Will assess change in knowledge and positive attitudes about risks, benefits, processes, and cultural factors associated with living kidney donation over time, and their associations with participant characteristics (i.e., age, literacy).

SECONDARY OUTCOMES:
Website use and satisfaction | 3 weeks
  Will assess satisfaction and use of website 3 weeks after enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Gordon, PhD, MPH, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - University of California, Davis, Davis, California
  - Northwestern Memorial Hospital (NMH), Chicago, Illinois

REFERENCES:
- [Derived] Gordon EJ, Feinglass J, Carney P, Vera K, Olivero M, Black A, O'Connor K, MacLean J, Nichols S, Sageshima J, Preczewski L, Caicedo JC. A Culturally Targeted Website for Hispanics/Latinos About Living Kidney Donation and Transplantation: A Randomized Controlled Trial of Increased Knowledge. Transplantation. 2016 May;100(5):1149-60. doi: 10.1097/TP.0000000000000932. PMID 26444846